CLINICAL TRIAL: NCT01307878
Title: Pre-operation Chemotherapy of Primary Tumor Resection for Colorectal Cancer Patients With Asymptomatic Resectable Primary Lesion and Synchronous Unresectable Liver-limited Metastases
Brief Title: New Adjuvant Chemotherapy of Asymptomatic Resectable Primary Lesion With Unresectable Liver-limited Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Ruijin Hospital (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xu jianmin, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECUT
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms; Chemotherapy; Maternal, Affecting Fetus
Keywords: Unresectable colorectal liver metastases; Pre-operation chemotherapy; Primary tumor resection; Survival
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm A (Experimental): Pre-PTR, chemotherapy regimen with either mFOLFOX6 plus cetuximab, bevacizumab or mFOLFOX6 alone were allocated, according the RAS genotype and patient affordability.
  Interventions: Drug: chemotherapy ± targeted therapy
- arm B (No Intervention): Upfront PTR, then chemotherapy regimen with either mFOLFOX6 plus cetuximab, bevacizumab or mFOLFOX6 alone were allocated, according the RAS genotype and patient affordability.

INTERVENTIONS:
Drug: chemotherapy ± targeted therapy — Chemotherapy regimen with either mFOLFOX6 plus cetuximab, bevacizumab or mFOLFOX6 alone were allocated, according the RAS genotype and patient affordability.
  Other Names: chemotherapy plus targeted therapy
  Arms: arm A

SUMMARY:
To evaluate the survival benefit of pre-operation chemotherapy of primary tumor tesection (PTR) compared upfront PTR for colorectal cancer (CRC) patients with an asymptomatic resectable primary tumor and synchronous unresectable liver-limited metastases with conversion therapy intent.

DETAILED DESCRIPTION:
Fast recovery with fewer postoperative complications, prevention of potential tumor-related complications during chemotherapy, life quality improvement, and also can alleviate the tumor load of patients, are some advantages of PTR that may play a role in improving cancer-specific survival. However, it should be pointed out that nearly all the retrospective and prospective studies for the beneficial of PTR enrolled more multi-organ metastases mCRC patients, and with palliative treatment purpose. As for unresectable colorectal liver-limited metastases (CRLMs) with good Eastern Cooperative Oncology Group performance status (ECOG PS), the primary objective is to make metastases resectable by high-intensity conversion therapy and achieved a state of no-evidence of disease. PTR were preferred performed before enrollment in some related RCT studies, including the CELIM study, CAIRO and CAIRO2 studies. Pooled-analysis of our two RCT studies, PTR pre or post chemotherapy for these unresectable liver-limited metastases patients had less morbidities and no mortalities, but no RCTs have focused on survival benefit of pre-operation chemotherapy of PTR for unresectable CRLMs.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 75 years old
* colorectal adenocarcinoma pathologically
* without any chemotherapy or radiotherapy
* unresectable liver metastasis and without other metastasis
* resectable colorectal cancer
* suitable for chemotherapy
* agreed by patients

Exclusion Criteria:

* age below 18 years old or greater than 75 years old
* haven't pathological diagnosis of colorectal adenocarcinoma
* with any chemotherapy or radiotherapy
* resectable liver metastasis or without other metastasis
* unresectable colorectal cancer
* unsuitable for chemotherapy
* not agreed by patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to 3 years
  Time from randomization to the date of disease progression or to death of any cause

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Time from randomization to death from any cause or the date of the last follow-up
Tumor response | Up to 6 months
  Response according to RECIST 1.1
Secondary resection rate Second radical resectability | Up to 6 months
  The rate of patients converted to resection for liver metastases
Surgical complications | 30 days after surgery
  The proportion of patients with any complications occurred within 30 days after surgery
Toxicity of chemotherapy | Up to 6 months
  Patients will be evaluated for Adverse Events at the start of each treatment cycle according to NCI CTC 3.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, Ph.D., M.D, Study Chair — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, Shanghai Municipality, China